CLINICAL TRIAL: NCT07087288
Title: The Effect of Artificial Intelligence Supported Case Analysis Method on Nursing Students' Knowledge, Case Management Performance and Nursing Diagnosis Determination Skills
Brief Title: Artificial Intelligence Supported Case Analysis and Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ayser DÖNER, Research Assistant, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Erciyessbfhem
Record Dates: First submitted 2025-07-09; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Nursing Students; Artificial Intelligence (AI)
Keywords: nursing student; airtificial intelligence; nursing education

STUDY DESIGN:
Intervention Model Description: In this study, nursing students were divided into three groups as traditional teaching group, case analysis group and artificial intelligence group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Traditional teaching group (No Intervention): The students in this group will be analysed by the responsible lecturer of the course.
- Case Analysis Group (Active Comparator): Students in this group will present the case of their choice from the clinic.
  Interventions: Other: Case Analysis
- Artificial Intelligence Group (Experimental): Students in this group will take artificial intelligence supported case analysis course.
  Interventions: Other: AI-supported case

INTERVENTIONS:
Other: AI-supported case — In the artificial intelligence supported case analysis course, students will listen to the audio video prepared by artificial intelligence.
  Arms: Artificial Intelligence Group
Other: Case Analysis — The case analysis will be made through the presentation prepared by the students in the group.
  Arms: Case Analysis Group

SUMMARY:
In this study, it was aimed to evaluate the effect of artificial intelligence-supported case analysis method on nursing students' knowledge, case management performances and nursing diagnosis determination skills.This study was conducted in a single-blind randomised controlled trial design. Students were randomly assigned to the traditional teaching group, the case analysis group and the artificial intelligence group.

DETAILED DESCRIPTION:
Background: In recent years, the integration of artificial intelligence technology into nursing education has been increasing.

Objective: In this study, it was aimed to evaluate the effect of artificial intelligence-supported case analysis method on nursing students' knowledge, case management performances and nursing diagnosis determination skills.

Design: This study was conducted in a single-blind randomised controlled trial design.

Method: The study was planned to include 107 students actively enrolled in the 4th grade Integrated Health Practices III course in the spring semester of the 2024-2025 academic year in the nursing department.Students were randomly assigned to the traditional teaching group, the case analysis group and the artificial intelligence group.Information form, Mentimeter application to determine the ability to determine nursing diagnoses and case management performance evaluation, and Quizizz application for knowledge test were used for data collection.In addition, a semi-structured interview form was used.

ELIGIBILITY:
Inclusion Criteria:

* Active fourth year nursing students in the spring term of the 2024-2025 academic year in which the study was conducted,
* Having taken the nursing process theoretical course before,
* Having a mobile phone with an internet connection,
* Students who have previously prepared a care plan specific to their inpatients in at least one internal medicine clinic

Exclusion Criteria:

* Students who do not take the Integrated Health Practices III course,
* Have not planned care for inpatients in internal medicine clinics in previous clinical practice,
* Students who did not agree to participate in the study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Case Management Performance | 3 hours
  In this study, nursing students' interest, focus, satisfaction and motivation levels in the evaluation of traditional teaching method, case analysis method and artificial intelligence supported case analysis method courses were evaluated with Visual Analogue Scale (VAS) over 10 points using Mentimeter application.
Nursing Diagnosis Determination Skills | 3 hours
  With the Mentimeter application, students were asked to identify 5 prioritised nursing diagnoses related to the case. There is no scoring here, but the application creates a word cloud where the most common answer is shown in a larger font.

CONTACTS AND LOCATIONS:
Overall Officials: AYSER DÖNER, Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Only a short protocol can be shared with other researchers.